CLINICAL TRIAL: NCT04061096
Title: Effectiveness Of Local Anesthesia In Molar Teeth With Molar Incisor Hypomineralization-A Prospective Study
Brief Title: Local Anesthesia in Molar Teeth With Molar Incisor Hypomineralization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Didem Sakaryali (Other)
Responsible Party: Sponsor-Investigator, Didem Sakaryali, Asst. Prof. Dr., Baskent University
Organization: Baskent University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Didem Sakaryali
Record Dates: First submitted 2019-08-10; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Anesthesia; Cold test; Electrical pulp test
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Masking Description: no need
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MIH-effected carious first permanent molar teeth (Active Comparator): MIH-effected carious permanent first molar teeth were well-demarcated white/yellow or brown/yellow enamel opacities which is a sign for hypomineralization and asymptomatic which meant to be without any spontaneous pain or pain during eating or drinking, percussion or palpation tenderness, formation of abcess or fistula.
  Interventions: Diagnostic Test: Evaluation of cold test; Diagnostic Test: Evaluation of electrical pulp test; Diagnostic Test: Evaluation of pain during the treatment
- not MIH-effected carious first permanent molar teeth (Active Comparator): The carious not MIH-effected teeth were only carious without any hypomineralize areas and asymptomatic which meant to be without any spontaneous pain or pain during eating or drinking, percussion or palpation tenderness, formation of abcess or fistula.
  Interventions: Diagnostic Test: Evaluation of cold test; Diagnostic Test: Evaluation of electrical pulp test; Diagnostic Test: Evaluation of pain during the treatment
- MIH-effected non-carious first permanent molar teeth (Placebo Comparator): MIH-effected teeth were carious permanent first molar teeth with well-demarcated white/yellow or brown/yellow enamel opacities which is a sign for hypomineralization and did not have any sign of caries.
  Interventions: Diagnostic Test: Evaluation of cold test; Diagnostic Test: Evaluation of electrical pulp test; Diagnostic Test: Evaluation of pain during the treatment
- not MIH-effected non-carious first permanent molar teeth (Placebo Comparator): not any signs of being caries or hypomineralization.
  Interventions: Diagnostic Test: Evaluation of cold test; Diagnostic Test: Evaluation of electrical pulp test; Diagnostic Test: Evaluation of pain during the treatment

INTERVENTIONS:
Diagnostic Test: Evaluation of cold test — Cold test evaluation to describe the sensitivity level of teeth due to induce the hydrodynamic forces in dentine tubules.
Diagnostic Test: Evaluation of electrical pulp test — Electrical pulp test evaluation to describe the sensitivity level of teeth due to induce the nerve fibers in pulp tissue.
Diagnostic Test: Evaluation of pain during the treatment — Describe the sensitivity level due to induce the hydrodynamic forces during treatment procedure.

SUMMARY:
To compare responses to electrical pulp test (EPT) and cold test among molar incisor hypomineralization (MIH)-effected and not MIH-effected carious teeth before and after administration of local anesthesia for caries removal.

DETAILED DESCRIPTION:
Fifty carious permanent first molar teeth (25 MIH-effected, 25 not MIH-effected) were included. Firstly, radiographic caries depth, International Caries Detection and Assessment System (ICDAS) codes and MIH levels of teeth were recorded. Then, during the treatment, EPT and cold test were performed before and after the administration of local anesthesia. Visual Analog Scale for Pain was used to evaluate cold test and pain during treatment. When interpreting results, significancy level was stated for the values of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants

Exclusion Criteria:

* Not being cooperative during treatment procedure

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Cold test results | Time frame of cold test evaluation was aproximately 1 hour for each participant.
  Visual Analog Scale for Pain was used to evaluate the cold tests for before and after the local anesthesia. Visual analog scale was used to rate the sensitivity level of patients with 6 different faces representing different levels of pain from "0=no pain" to "10=unbearable pain".
Electrical pulp test results | Time frame of electrical pulp test evaluation was aproximately 1 hour for each participant.
  Electrical pulp test values at which patients felt sensitive were recorded.
Pain during the treatment | Pain during the treatment was evaluated for aproximately 1 hour for each participant.
  Visual Analog Scale for Pain was used to evaluate the pain during the treatment. Visual analog scale was used to rate the sensitivity level of patients with 6 different faces representing different levels of pain from "0=no pain" to "10=unbearable pain".

CONTACTS AND LOCATIONS:
Overall Officials: Didem Sakaryali, Asst.Prof., Principal Investigator — Baskent University

IPD SHARING:
Plan to Share IPD: No
The authors decided to share the information of this study after the study will be published in a scientific journal.